CLINICAL TRIAL: NCT00448344
Title: Family-Supported Smoking Cessation for Chronically Ill Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 05-202
Record Dates: First submitted 2007-03-14; First posted 2007-03-16 (Estimated); Results first posted 2014-08-27 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Disease; Neoplasm; Cardiovascular Disease; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus; Hypertension
Keywords: veterans; smoking cessation
MeSH Terms: conditions — Chronic Disease; Neoplasms; Cardiovascular Diseases; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus; Hypertension; Smoking Cessation | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Family-supported smoking cessation
  Interventions: Behavioral: Family-supported
- Arm 2 (Other): Standard smoking cessation
  Interventions: Behavioral: Standard Telephone counseling

INTERVENTIONS:
Behavioral: Family-supported — Group receives quit kit, option for nicotine replacement therapy, and 5 telephone counseling sessions with the goal of attaining social support during the process of quitting smoking
  Other Names: Intervention
  Arms: Arm 1
Behavioral: Standard Telephone counseling — Group receives quit kit, option for nicotine replacement therapy, and 5 standard smoking cessation telephone counseling sessions
  Other Names: Control
  Arms: Arm 2

SUMMARY:
The overarching aim of the study is to evaluate in a randomized trial the impact of a family-supported intervention compared to a standard veteran-focused telephone counseling control group to promote smoking cessation among cancer and heart disease patients.

DETAILED DESCRIPTION:
ANTICIPATED IMPACT(S) ON VETERAN'S HEALTHCARE:

Veterans with chronic disease who continue to smoke exact a significant burden on the VA health care system. Effective smoking cessation programs, that target veterans who continue to smoke after the diagnosis of a smoking-related chronic illness, are needed.

BACKGROUND/RATIONALE:

Chronic diseases related to tobacco exposure are common among veterans. Persistent tobacco use after being diagnosed with these diseases decreases quality of life and survival. Yet, 30% of veterans with these conditions continue to smoke. Researchers have found that the social environment is important for smokers. In our current NCI-funded study, 70% of veterans with lung cancer identified at least one family member who smokes and 45% live with a family member that smokes. A family-supported smoking cessation intervention timed to follow a veteran's diagnosis of cancer or heart disease could be effective for helping veterans quit smoking.

OBJECTIVES:

The overarching aim of the study is to evaluate in a randomized trial the impact of a family-supported intervention compared to a standard veteran-focused telephone counseling control group to promote smoking cessation among cancer and heart disease patients.

AIM 1: To evaluate the impact of a family-supported intervention on rates of abstinence from cigarettes (self-reported 7-day point prevalent abstinence) at 2 weeks, and 12-month post-treatment follow-ups.

Hypothesis 1: Abstinence rates will be significantly higher among veterans who receive the family-supported intervention than those who receive the standard telephone counseling control.

AIM 2: To evaluate the impact of a family-supported intervention on perceived support for quitting 2 weeks and 12-month post-treatment follow-ups.

Hypothesis 2: Perceived support for quitting smoking will be significantly greater among veterans who receive the family-supported intervention than those who receive the standard telephone counseling control.

AIM 3: To measure the impact of a family-supported intervention on quality of life in veterans 2 weeks, and 12-month post-treatment follow-ups.

Hypothesis 3: Symptom-related quality of life will be significantly greater among veterans who receive the family-supported intervention than those who receive the standard telephone counseling control.

METHODS: Proposed is a two-group design in which 470 veterans who smoke will be randomized to receive:

STANDARD TELEPHONE COUNSELING control including a letter from a VA physician encouraging the patient to quit smoking, nicotine replacement (if not contraindicated), a self-help cessation kit, and 5 standard telephone counseling calls; or FAMILY-SUPPORTED intervention that includes all components of the control arm plus a Family-supported intervention that includes a support skills booklet and an additional telephone counseling protocol focusing on social support. .

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Durham VA for ongoing care
* Seen at a DVAMC clinic for care of cancer or cardiovascular disease within the previous 3 months
* Current smokers and planning to quit smoking in the next 30 days

Exclusion Criteria:

* Active diagnosis of psychosis documented in medical record
* Does not have access to a telephone
* Refusal to provide informed consent
* Severely impaired hearing or speech

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2008-02; Primary Completion 2010-09 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Anne Bastian, MD MPH, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

REFERENCES:
- [Result] Bastian LA. If it is as simple as AAAAA B C, why don't we do it? J Gen Intern Med. 2009 Feb;24(2):284-5. doi: 10.1007/s11606-008-0896-2. No abstract available. PMID 19139966
- [Result] Bastian LA, Sherman SE. Effects of the wars on smoking among veterans. J Gen Intern Med. 2010 Feb;25(2):102-3. doi: 10.1007/s11606-009-1224-1. No abstract available. PMID 20077050
- [Result] Rohrer LD, Gierisch JM, Fish LJ, Blakeney JK, Bastian LA. A five-step guide for moving from observational studies to interventional research for women veterans. Womens Health Issues. 2011 Jul-Aug;21(4 Suppl):S98-102. doi: 10.1016/j.whi.2011.05.004. No abstract available. PMID 21724150
- [Result] Fish LJ, Gierisch JM, Stechuchak KM, Grambow SC, Rohrer LD, Bastian LA. Correlates of expected positive and negative support for smoking cessation among a sample of chronically ill veterans. Addict Behav. 2012 Jan;37(1):135-8. doi: 10.1016/j.addbeh.2011.08.013. Epub 2011 Sep 17. PMID 21978930
- [Result] Bastian LA, Fish LJ, Gierisch JM, Rohrer LD, Stechuchak KM, Grambow SC. Comparative effectiveness trial of family-supported smoking cessation intervention versus standard telephone counseling for chronically ill veterans using proactive recruitment. Comparative Effectiveness Research. 2012 Jan 1; 2012(2):45-56.
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Bastian LA, Fish LJ, Gierisch JM, Stechuchak KM, Grambow SC, Keefe FJ. Impact of Smoking Cessation on Subsequent Pain Intensity Among Chronically Ill Veterans Enrolled in a Smoking Cessation Trial. J Pain Symptom Manage. 2015 Dec;50(6):822-9. doi: 10.1016/j.jpainsymman.2015.06.012. Epub 2015 Jul 22. PMID 26210348

RESULTS

PARTICIPANT FLOW:
Groups:
- Family-supported Smoking Cessation: Family-supported smoking cessation
  Family-supported: Group receives quit kit, option for nicotine replacement therapy, and 5 telephone counseling sessions with the goal of attaining social support during the process of quitting smoking
- Standard Smoking Cessation: Standard smoking cessation
  Standard Telephone counseling: Group receives quit kit, option for nicotine replacement therapy, and 5 standard smoking cessation telephone counseling sessions
Period: Overall Study
Arm/Group | Family-supported Smoking Cessation | Standard Smoking Cessation
Started | 235 | 236
Completed | 205 | 200
Not Completed | 30 | 36
Not completed — Lost to Follow-up | 20 | 22
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Death | 3 | 4
Not completed — Physician Decision | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 235 | 236 | 471
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (8) | 59.2 (7.7) | 59.2 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 214 | 217 | 431
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 7 | 11
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 92 | 96 | 188
  White | 130 | 121 | 251
  More than one race | 8 | 7 | 15
  Unknown or Not Reported | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Impact of a Family-supported Intervention on Rates of Abstinence From Cigarettes Compared to a Standard Intervention
Description: self-reported 7-day point prevalent abstinence
Time Frame: 5 months
Measure: Number; unit: percentage of participants that quit
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 235 | 236
percentage of participants that quit | 19.8 | 22.0

2. Secondary Outcome: The Impact of a Family-supported Intervention on Abstinence at 12-month Follow-up
Description: self-reported 7- day point prevalent abstinence
Time Frame: 12-months follow-up
Measure: Number; unit: percentage of participants that quit
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 235 | 236
percentage of participants that quit | 22.4 | 22.4

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 7/235 | 13/236
Other Adverse Events (participants affected / at risk) | 0/235 | 0/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=235) | Arm 2 (N=236)
deceased during study (Cardiac disorders) | 7 | 13 — not related to study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes